CLINICAL TRIAL: NCT03518749
Title: Effects of tDCS-enhanced Cognitive Control Training on Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 01EE1403D-2
Record Dates: First submitted 2018-04-13; First posted 2018-05-08 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Depression Unipolar
Keywords: Depression; transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1mA anodal tDCS + cognitive control training (Active Comparator): 1 mA anodal tDCS will be administered to the left dlPFC (F3) for 23 mins during the performance of a cognitive control training.
  Interventions: Other: 1mA tDCS; Behavioral: Cognitive control training
- 2mA tDCS + cognitive control training (Active Comparator): 2 mA anodal tDCS will be administered to the left dlPFC (F3) for 23 mins during the performance of a cognitive control training.
  Interventions: Other: 2mA tDCS; Behavioral: Cognitive control training
- sham tDCS + cognitive control training (Placebo Comparator): Sham tDCS (30 secs of tDCS) will be administered to the left dlPFC (F3) with 2mA at the beginning of a cognitive control training.
  Interventions: Behavioral: Cognitive control training

INTERVENTIONS:
Other: 1mA tDCS — transcranial direct current stimulation with the intensity of 1mA
  Arms: 1mA anodal tDCS + cognitive control training
Other: 2mA tDCS — transcranial direct current stimulation with the intensity of 2mA
  Arms: 2mA tDCS + cognitive control training
Behavioral: Cognitive control training — cognitive control training with the PASAT

SUMMARY:
Deficient cognitive control (CC) is one of the central characteristics of major depression (MD). Hypoactivation of the dorsolateral prefrontal cortex (dlPFC) has been linked with this deficit. Antidepressants and cognitive-behavioral therapies modify CC most-likely as a common mechanism of treatment. Transcranial direct current stimulation (tDCS) is a safe, simple and effective non-invasive method to modulate the cortical excitability. It has been shown, that the activity of the dlPFC can be modulated by transcranial direct current stimulation (tDCS) with polarity-dependent learning-phase specific effects on performance that, when combined with training, can outlast the stimulation.

The goal of this randomized, sham-controlled, rater blind clinical trial is to investigate the effect of a tDCS-enhanced CC Training (CCT) on depressive symptom severity and compare the stimulation intensities 1mA, 2mA and sham tDCS. Overall, the study will include 57 participants (n = 19 per group). Each participant will complete 12 training sessions with online sham/ anodal tDCS.

As a training task we will use an adaptive version of the paced auditory serial addition task (PASAT). In the PASAT, digits are presented auditive and participants have to add the current digit to the digit they heard before. In the adaptive version the interstimulus-intervals decrease (increase) when four consecutive trials are correct (incorrect). The PASAT is known to elicit frustration. Participants have to exert cognitive control over these emotions to complete the task successfully.

Before, during and after the training symptom severity will be assessed. Baseline and post-training performance in the PASAT and in a transfer task (delayed working memory task, DWM) will be measured.

To further explore variables that influence the effect of tDCS on depressive symptom severity we will measure brain activity (EEG, NIRS), heart rate, global functioning (GAF), emotion regulation strategies, self-esteem, mood ratings and subjective performance ratings before and after the training and collect genetic factors.

Sustainability of the training effects will be measured at a follow-up visit (3 months later).

ELIGIBILITY:
Inclusion Criteria:

* current Major Depressive Episode
* right handedness

Exclusion Criteria:

* history of seizures
* Intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* pregnancy
* use of mood stabilizers
* diagnosed bipolar disorder
* current substance abuse (nicotine excluded)
* current substance addiction (nicotine excluded)
* diagnosed psychotic diseases
* diagnosed anorexia nervosa
* diagnosed personality disorders: cluster A, antisocial personality disorder,
* borderline personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of MADRS scores | Assessment one week before training start (week -1, day -5 on average) and in the last training session (week 4, day 26)
  Change in Depressive Symptom severity will be measured with the Montgomery-Åsberg Depression Rating Scale (MADRS) from Baseline session to the last stimulation session, scale range from 0 to 60 points, higher scores indicate a more severe depression

SECONDARY OUTCOMES:
BDI scores | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Beck Depression Inventory
Number of correct trials in the PASAT | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Performance in the PASAT. Number of correct trials.
RT in the DWM | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Reaction time in the transfer task, a delayed working memory task (DWM)
Number of correct trials in the DWM | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Number of correct trials in the transfer task, a delayed working memory task (DWM)
GAF score | Assessment one week before training start (week -1, day -5 on average) and in the post training session (week 5, day 31 on average)
  Global Assessment of Functioning
Delta Mood ratings | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Mood changes (PANAS delta) through the PASAT performance: the positive and negative affective schedule (PANAS) will be conducted immediately before and after the PASAT performance. The change in mood ratings (PANAS delta = PANAS pre PASAT - PANAS post PASAT) will be the outcome measure.
Subjective performance ratings | Assessment one week before training start (week -1, day -5 on average), in the post training session (week 5, day 31 on average) and at follow-up (week 17, day 110 on average)
  Participants will be asked to rate their performance and overall cognitive abilities on a likert scale.
Electroencephalography (EEG) measures | Assessment one week before training start (week -1, day -5 on average) and in the post training session (week 5, day 31 on average)
  EEG will be conducted to measure resting state oscillations and event related potentials stimulus locked to the presented feedback in the PASAT
Prefrontal Brain activity (NIRS) | Assessment one week before training start (week -1, day -5 on average) and in the post training session (week 5, day 31 on average)
  Functional Near Infrared Spectroscopy will be used to measure frontal brain activity: resting state and during task performance.
Course of MADRS scores | Assessment once a week during training (week 1, 2 and 3 at day 5, 12 and 19 respectively on average) and at the follow up visits (week 5 and 17, day 31 and 110 on average)
  Depressive Symptom severity will be measured with the Montgomery-Åsberg Depression Rating Scale
Prefrontal Brain activity (NIRS) as a predictor | Assessment one week before training start (week -1, day -5 on average)
  The investigators will analyze if frontal brain activity measured with NIRS during resting state and task performance can contribute to the prediction of the effectiveness of the tDCS training.
Electroencephalography (EEG) measures as a predictor | Assessment one week before training start (week -1, day -5 on average)
  The investigators will analyze if resting state oscillations and event related potentials stimulus locked to the presented feedback in the PASAT can contribute to the prediction of the effectiveness of the tDCS training.
Genetic factors as predictors | Assessment one week before training start (week -1, day -5 on average)
  The investigators will analyze if genetic factors involved in neuroplasticity (5-HTTLPR, BDNF, COMT) can contribute to the prediction of the effectiveness of the tDCS training.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sommer A, Fallgatter AJ, Plewnia C. Investigating mechanisms of cognitive control training: neural signatures of PASAT performance in depressed patients. J Neural Transm (Vienna). 2022 Jun;129(5-6):649-659. doi: 10.1007/s00702-021-02444-7. Epub 2021 Nov 23. PMID 34812928